CLINICAL TRIAL: NCT06446219
Title: A Retrospective Analysis of the Efficacy and Safety Comparison of Upadacitinib and Vedolizumab in Second-line Treatment for Crohn's Disease
Brief Title: Efficacy and Safety Comparison of Upadacitinib and Vedolizumab in Second-line Treatment for Crohn's Disease
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024ZSLYEC-257
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Upadacitinib(UPA): Upadacitinib, a selective Janus kinase (JAK) inhibitor taken orally, is being assessed for its unique capacity to attenuate inflammatory pathways in Crohn's Disease at a cellular level by selectively inhibiting Janus kinase(JAK)1, a pathway integral to inflammatory cytokine production. This study focuses on its use as main therapy for Chinese patients unresponsive to conventional Crohn's Disease treatments, such as tumor necrosis factor-α inhibitor. Rinvoq is the marketed drugs for clinical use, whose oral dosage is 45 mg per day during the induction period and 15 mg/30 mg per day during maintenance period, and the induction period would last for 8 weeks.
- Vedolizumab(VDZ): Vedolizumab, a monoclonal antibody targeting integrin α4β7, is used to inhibit recruitment of inflammatory cells. This drug is always used as second-line treatment for patients with moderate-to-severe active stage Crohn's Disease who fail to respond to conventional treatments such as tumor necrosis factor-α inhibitor. This study uses Vedolizumab as control group to illustrate the efficacy and safety of Upadacitinib in second-line treatment for Crohn's Disease. Entyvio is the marketed drugs for clinical use, should be given intra-arterially in week 0, 2, 6 and every subsequent 8 weeks.

SUMMARY:
This study focuses on Upadacitinib, a new oral and small-molecular medication that inhibits specific enzymes involved in inflammation. The goal is to determine efficacy and safety of Upadacitinib for Crohn's Disease patients in China compared with Vedolizumab, which is used to inhibit recruitment of inflammatory cells. Crohn's Disease significantly affects individuals' quality of life and imposes a high burden on society and healthcare systems. Current treatments don't work for everyone, and some patients may need surgery. Upadacitinib has shown promise in other countries for treating Crohn's Disease and related conditions, and has been approved by the US FDA for such use.

The investigators' retrospective and multicenter study looks back at patient records from multiple hospitals to analyze the outcomes of those who have received Upadacitinib and Vedolizumab. Investigators aim to enroll patients treated between January 2020 and March 2024, who received follow-up for more than 12 weeks. For patients, families, and healthcare providers, this research could provide a potential new treatment option for Crohn's Disease. Better efficacy and safety of Upadacitinib than Vedolizumab could lead to better management of the disease, possibly reducing the need for surgery and improving the quality of life. The ultimate goal is to provide more personalized and effective treatment strategies for Crohn's Disease patients in China.

DETAILED DESCRIPTION:
This retrospective, multicenter study is designed to compare the efficacy and safety of Upadacitinib and Vedolizumab in second-line treatment for Crohn's Disease, the former is an oral selective enzyme inhibitor, and the latter is a monoclonal antibody targeting integrin α4β7. Crohn's Disease poses a significant impact on the quality of life for individuals and presents a considerable challenge to healthcare systems due to the societal burdens it incurs. While current therapeutic interventions offer relief, these interventions fail to suffice for all patients, with some requiring surgical intervention. Despite the approval of Upadacitinib by the US FDA and its promising application in other nations for Crohn's Disease management, there is a scarcity of data on its effectiveness and safety among Chinese patients. The investigators' research aims to fill this knowledge gap by retrospectively analyzing patient records from multiple hospitals across China. The study targets the adult patients that has received follow-up for more than 12 weeks between January 2020 and March 2024. By assessing the outcomes of these patients, the investigators' objective is to ascertain the potential of Upadacitinib as a viable treatment alternative, which may revolutionize the current Crohn's Disease treatment paradigm in China.The implications of this study are significant for patients, their families, and healthcare providers, as it could herald a new therapeutic avenue for Crohn's Disease management. A clearer understanding of Upadacitinib's role in disease control could enhance patient care by decreasing the necessity for surgical procedures and ameliorating life quality for Crohn's Disease sufferers. The overarching ambition of this research is to pave the way for more individualized and efficacious treatment methodologies for the Crohn's Disease patient populace in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were hospitalized in our institution or its branches between January 2020 and March 2024.
* Patients aged 18 years or older.
* Confirmed as moderately-to-severely active Crohn's disease according to Chinese clinical practice guideline on the management of Crohn's disease (2023,Guangzhou).
* Failure to respond to or tolerate anti-tumor necrosis factor-α inhibitors (Infliximab, Adalimumab).
* Follow-up time for no less than 12 weeks.

Exclusion Criteria:

* Patients who have previously used Upadacitinib and Vedolizumab.
* With insufficient clinical data at baseline, 12 weeks in the Upadacitinib group and 14 weeks in the Vedolizumab group to evaluate the efficacy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients aged 18 and older who were hospitalized for Crohn's Disease between January 2020 and March 2024 at our institution or its branches, and who have been received follow-up for no less than 12 weeks prior to March 2024. The study population should also failure to respond to or tolerate anti-tumor necrosis factor-α inhibitors (Infliximab, Adalimumab). The focus is on adults with a confirmed diagnosis to assess the efficacy in inducing clinical remission and altering disease progression. Exclusion criteria include unclear diagnosis, patients under 18, previously using Upadacitinib/Vedolizumab and absence of clinical data, ensuring a uniform group for valid results.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Steroid-Free Clinical Remission | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  Steroid-Free Clinical Remission in Crohn's Disease is defined as a Crohn's disease activity index(CDAI) score of less than 150, achieved without the use of corticosteroids.

SECONDARY OUTCOMES:
Clinical Remission | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  Clinical Remission in Crohn's Disease is defined as a Crohn's disease activity index(CDAI) score of less than 150
Clinical Response | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  Clinical Response in Crohn's Disease is a decrease in Crohn's disease activity index(CDAI) score by 70 points or more from baseline.
Endoscopic Remission | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  A simple endoscopic score for Crohn's disease(SES-CD) score of 2 or less indicates endoscopic remission
Endoscopic Response | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  Endoscopic Response in Crohn's Disease is a decrease in simple endoscopic score for Crohn's disease(SES-CD) score by 50 percent or more from baseline.
Mucosal Healing | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  A simple endoscopic score for Crohn's disease(SES-CD) score of 0 is indicative of mucosal healing
Radiological Remission | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  Defined as the complete disappearance or minimization of intestinal inflammation on imaging studies, signifying no visible lesions, normalized wall thickness, absence of strictures or obstructions, and no new areas of disease. Radiographic remission is an important indicator of deep remission in disease treatment goals.
Radiological Response | Upadacitinib group: assessed at 12 weeks; Vedolizumab group: assessed at 14 weeks;
  Typically defined as a significant reduction in the size of affected areas, decreased wall thickness, and decreased markers of inflammation observed through imaging methods such as MRI or CT scans. A radiographic response indicates a reduction in disease activity but may not represent complete disease remission.

CONTACTS AND LOCATIONS:
Locations (1):
- the Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No